CLINICAL TRIAL: NCT05242016
Title: The Effect of Structured Individiual Reminiscence on Symptom Management, Life Satisfaction and Self Transcendence of Palliative Care Patients
Brief Title: Structured Individiual Reminiscence on Self Transcendence of Palliative Care Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bandırma Onyedi Eylül University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Canan BOZKURT, Research Assistant, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: bandirma
Record Dates: First submitted 2022-01-02; First posted 2022-02-16 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Palliative Care
Keywords: self-transcendence; structured reminiscence; life satisfaction; symptom management; palliative care; well-being
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Questionnaires are administered to three groups: structured individual reminiscence, unstructured social interview, and control, before the application (day 1) and after the application (day 15).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- structured individual reminiscence (Experimental): Sessions, in chronological order; Starting with birth, it is planned to progress through life years by focusing on important events. In the sessions, considering the age and individual characteristics of the patients, the house and region where they were born and raised, childhood and school memories, childhood and school friends, youth years and friends, business life, if any, marriage process, birth of the first child, happy memories about children, successful events, old holidays It is talked about subjects such as unforgettable people or events, happy places to visit, old meals, old items, old songs. In each session, different sensory stimuli (visual, auditory, tactile, smelling, tasting) are used according to the subject.
  Interventions: Other: structured individual reminiscence
- unstructured social interview (Placebo Comparator): Unstructured social interviews are conducted on topics such as current events not related to recollection, information specific to the individual patient wants to share, illness/diseases, hobbies, and activities.
  Interventions: Other: unstructured social interview
- Control (No Intervention): There is no intervention other than standard nursing care.

INTERVENTIONS:
Other: structured individual reminiscence — reminiscence therapy
  Arms: structured individual reminiscence
Other: unstructured social interview — placebo
  Arms: unstructured social interview

SUMMARY:
Palliative Care is the care offered by a simultaneous multidisciplinary approach with all treatments aimed at preventing/alleviating suffering and increasing the quality of life by early identifying all physical, psycho-social and spiritual needs, especially pain, to individuals and their families who face problems arising from life-threatening diseases. philosophy. For this reason, it includes the quality of life and the positive effect of the disease process. Symptom management starts from the moment of diagnosis and lasts until the moment of death, and as in all areas, complementary therapies are very important in palliative care as well as pharmacological treatment.

DETAILED DESCRIPTION:
It is thought that increasing the quality of life of palliative care patients, making sense of the past life and transforming the negative perspective into a positive one, as well as the symptoms seen in the process until death, can contribute positively to the quality of life of the individual. The reason for this is personality development, which he mentioned in the Psychosocial Development Theory, which was introduced in the 1950s. He reported that personality development lasts for a lifetime and consists of eight stages, and the last stage will be hopeless in an individual whose self-integrity is not complete. Because, according to the theory, every individual has accepted all the experiences he has lived in his life as they are, assimilated and adapted to complete the integrity of the self. In this totality, there is no regret for the past, no fear and anxiety for the future. Despair will cause the individual to experience fear of death because death is an inevitable end and should be expected in peace as a natural part of life. Based on this theory, a gerontologist and psychiatrist argued in his 1963 study Life Review that the act of reviewing the past is about integrating and interpreting experiences in the dimension of analyzing the past. After the word reminiscence was derived, studies emerged as Reminiscence Therapy by structuring the review process of life. Although it originally emerged as a psychoanalytic concept, reminiscence therapy has been used as a component of nursing in long-term care settings. Nurses began using Reminiscence Therapy in the late 1960s and published their experiences in the 1970s. At that time, the purpose of nurses in applying Reminiscence Therapy was to help older individuals reframe their experiences and prepare for death. In 1978, a nurse described some of the therapeutic factors of Reminiscence Therapy as identification, socialization, intergenerational sharing, memory stimulation, and self-actualization. As a definition of self-transcendence, it was first defined in British literature by Maslow in 1969 as the highest, most inclusive or holistic consciousness that transcends time, culture and self. Later, Maslow modified the "Hierarchy of Needs" model and reported adding self-actualization as a motivational step. Over time, a middle-class nursing theory named "Self-Transcendence Theory" was developed by Pamela G. Reed (1991). Nursing as a science is thought to be based on the self-transcendence theory developed by Pamela G. Reed for the nursing care they will apply to palliative care patients in a conceptual framework. Because in his theory, Reed argues that individuals who experience chronic illness, loss and aging or who accompany others with these events should face vulnerability. It has been reported that nurses can facilitate the individual's self-transcendence and support the welfare potential of individuals. Meditation, prayer, visualization, life review, structured reminiscence, self-reflection, and journaling are techniques of self-transcendence that nurses can facilitate to help their patients recognize their own patterns of healing. In the light of this information, the aim of this study is to investigate the effect of structured individual reminiscence on symptom management, life satisfaction and self-transcendence of palliative care subordinates.

ELIGIBILITY:
Inclusion Criteria:

* Speaking and understanding Turkish
* Those who volunteered to participate in the research
* Inpatient in Palliative Care Service
* Without clinical diagnosis of dementia, cognitive impairment, agitation and delirium
* No hearing or vision problems

Exclusion Criteria:

* Patients who are planned to be transferred and/or discharged to another unit/institution within the estimated period of investigation (15 days) by the physician and who do not have a life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-05-25 (Estimated)

PRIMARY OUTCOMES:
self-transcendence scale | 15 days
  The change in self-transcendence scores of the patients in the structured individual reminiscence group after the application compared to the pre-application. The self-transcendence scale score ranges from 15 to 60, and an increase in scores indicates that the individual is self-actualizing.
life satisfaction | 15 days
  The change life satisfaction in scores of the patients in the structured individual reminiscence group after the application compared to the pre-application. The life satisfaction scale score ranges from 5-35, and an increase in the score indicates that the individual's life satisfaction is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandirma Training and Research Hospital, Bandırma, Balikesi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bozkurt C, Yildirim Y. The effectiveness of reminiscence therapy on the symptom management, the life satisfaction, and the self-transcendence in palliative care patients: a randomized controlled trial. Support Care Cancer. 2024 Jun 14;32(7):431. doi: 10.1007/s00520-024-08626-9. PMID 38874763

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT05242016/SAP_000.pdf